CLINICAL TRIAL: NCT03917134
Title: Efficacy of the Use of Metronidazole After Laparoscopic Hysterectomy for the Prevention of Vaginal Cellulitis or Vaginal Cuff Abscess. Multicentric Triple-blind Randomized Controlled Trial
Brief Title: Prevention of Vaginal Cellulitis or Vaginal Cuff Abscess After Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CES University (Other)
Collaborators: Lafrancol S.A. (Industry); Prolab S.A (Unknown); Clínica del prado (Unknown); Clínica comfamiliar pereira (Unknown)
Responsible Party: Principal Investigator, Claudia López, Principal investigator, CES University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 815
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hysterectomy; Cellulitis; Vaginosis; Abscess; Cuff
MeSH Terms: conditions — Cellulitis; Vaginal Diseases; Abscess | interventions — Cephalosporins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cephalosporin + Metronidazole (Experimental): In this arm, patients randomly selected, will receive cephalosporin in doses of 2 grams administered intravenously before surgery. metronidazole vaginal ovules of 500mg twice a day for 5 days after surgery
  Interventions: Drug: cephalosporin + Metronidazole Vaginal
- cephalosporin + placebo (Placebo Comparator): In this arm, patients randomly selected, will receive cephalosporin in doses of 2 grams administered intravenously before surgery. placebo vaginal ovules twice a day for 5 days after surgery
  Interventions: Drug: cephalosporin + Placebos

INTERVENTIONS:
Drug: cephalosporin + Metronidazole Vaginal — administration of cephalosporin in doses of 2 grams administered intravenously before surgery and metronidazole vaginal ovules 500mg twice a day for 5 days after performing laparoscopic hysterectomy
  Arms: cephalosporin + Metronidazole
Drug: cephalosporin + Placebos — administration of cephalosporin in doses of 2 grams administered intravenously before surgery and vaginal ovules of placebo twice a day for 5 days after performing laparoscopic hysterectomy
  Arms: cephalosporin + placebo

SUMMARY:
Operative site infection remains the most common complication after performing a gynecological procedure, and has a great implication in the morbidity and mortality of patients. Gynecological procedures, including laparoscopic hysterectomy, represent a unique challenge due to the amount of microorganisms found at the skin level of the vagina or the endocervix.

However, there is no clear evidence that the complication decreases with the use of postoperative antibiotics.

With the completion of this study, a multicentre triple-blind controlled randomized controlled trial is intended to determine the behavior of the application of this intervention.

Patients who attend an outpatient clinic with benign pathology will be selected, in which indication of laparoscopic hysterectomy, consents are completed and research content is widely explained. Prior to surgery, the sample is taken for a gram of vaginal discharge and in the post-surgical phase delivery of the medication will be performed. Follow-up will be carried out by surgical control and by telephone.

The investigator intend to find that with the prophylaxis not only of presurgical cephalosporin, but with the formulation of metronidazole ovules in the postoperative, the incidence of laparoscopic post-hysterectomy vaginal abscess and cellulitis of cuff is reduced.

DETAILED DESCRIPTION:
The development of the project will be carried out in the facilities of the Prado clinic in the city of Medellín and the Comfamily Clinic in the city of Pereira. Initially to the participants who attend by external consultation for assessment by the laparoscopic gynecology group that are candidates to perform a laparoscopic hysterectomy, they will be given general information about the research in development and its possible participation. Later on the day of surgery in the preparation room and before receiving any medication, The assigned investigator as assistant to the surgery will explain in detail the protocol of the investigation, the commitments acquired by the participant and the possibilities of withdrawal of the same, you will obtain the signature and trace of the informed consent. With the aim of not delaying the 7 am surgical program, a weekly resident will be assigned to inform and fill out the forms of the first patients scheduled for hysterectomy.

Advance by means of a table of random numbers generated in EPIDAT and that is hidden for the researcher. Participants will be assigned to one of the 2 groups, the intervention group will receive the treatment scheme with metronidazole 500mg ovules every 12 hours for 5 days and the control group will receive a placebo.

After this in the surgery room and with the participants under general anesthesia, the sample will be taken for gram of vaginal discharge, previous marking of the plate, with the initials of names and surnames and the patient's identification number, With the use of a speculum and applicator the sample will be taken in the sack bottoms or vaginal walls, which will be sent to the Prolab laboratory in the city of Medellín and the laboratory of the Comfamily clinic in the city of Pereira. for its processing, standardization will be made prior to reading it with the staff of both laboratories.

For the diagnosis of bacterial vaginosis, the Nugent criteria will be used. In this method, the morphotypes corresponding to large Gram-positive bacilli, small Gram-negative bacilli and curved variable Gram bacilli are quantified. And a value is assigned according to the findings. The interpretation of the results is numerical based on the score obtained by adding the crosses of the morphotypes of the bacteria present in the vaginal discharge: 7 or more points are diagnostic of bacterial vaginosis, from 4 to 6 points is considered intermediate and from 0 to 3 is considered normal.

At the end of the surgical procedure, the investigator will complete the completion of Annex 1, will go to the pharmaceutical service where he will request the corresponding product to the patient. The pharmacy staff will verify the assigned number in the randomization table and deliver the medication and the resident will take it to the recovery room with its respective formula.

The assigned investigator will conduct a telephone interview 7 days after the procedure to assess the post-surgical evolution, will be questioned about the presence of symptoms that may be related to an infectious process. Between 10-15 days of the surgical procedure, the gynecologist will perform the post-surgical review in an outpatient clinic to assess the evolution of the patient and re-evaluate the result of the pathology. The Gram result of vaginal discharge, the pathology and the evolution note made by the surgeon will be reviewed with the aim of detecting any diagnosed complication. Finally, 30 days after the procedure, the last telephone follow-up will be performed to detect the presence of any infection. of the operative site.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 55 years old scheduled for laparoscopic hysterectomy for benign pathology in the two centers linked to the study (Clínica del Prado and Pereira community clinic), who have been informed of their participation in the study and who have signed informed consent.
* Patients who are able to communicate by telephone and answer questions

Exclusion Criteria:

* Patients who are participating in another study of antibiotic treatment.
* Patients who have a known allergy to imidazole medications.
* Patients with current diagnosis of bacterial vaginosis.
* Patients with current treatment or 30 days prior to surgery for bacterial vaginosis or antibiotic treatment for another pathology.
* Patients who do not reside in Medellín or in its nearby municipalities and can not attend the scheduled evaluation.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of cellulitis and vaginal cuff abscess | 30 days

SECONDARY OUTCOMES:
percentage of patients who will undergo laparoscopic hysterectomy have bacterial vaginosis at the time of the procedure. | 15 days
need to perform additional procedures as part of the treatment in each of the groups. | 30 days
percentage of patients who comply with the prescribed treatment completely. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA LOPEZ, Gynecologist, Principal Investigator — CES University - Clínica del prado
Locations (2):
- Colombia (2):
  - Clinica del prado, Medellín
  - Clínica comfamiliar pereira, Pereira

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] ACOG practice bulletin No. 104: antibiotic prophylaxis for gynecologic procedures. Obstet Gynecol. 2009 May;113(5):1180-1189. doi: 10.1097/AOG.0b013e3181a6d011. No abstract available. PMID 19384149
- [Result] Lowe NK, Neal JL, Ryan-Wenger NA. Accuracy of the clinical diagnosis of vaginitis compared with a DNA probe laboratory standard. Obstet Gynecol. 2009 Jan;113(1):89-95. doi: 10.1097/AOG.0b013e3181909f63. PMID 19104364
- [Result] Brachman PS, Dan BB, Haley RW, Hooton TM, Garner JS, Allen JR. Nosocomial surgical infections: incidence and cost. Surg Clin North Am. 1980 Feb;60(1):15-25. doi: 10.1016/s0039-6109(16)42030-x. PMID 7361218
- [Result] Persson E, Bergstrom M, Larsson PG, Moberg P, Platz-Christensen JJ, Schedvins K, Wolner-Hanssen P. Infections after hysterectomy. A prospective nation-wide Swedish study. The Study Group on Infectious Diseases in Obstetrics and Gynecology within the Swedish Society of Obstetrics and Gynecology. Acta Obstet Gynecol Scand. 1996 Sep;75(8):757-61. doi: 10.3109/00016349609065742. PMID 8906013
- [Result] Oduyebo OO, Anorlu RI, Ogunsola FT. The effects of antimicrobial therapy on bacterial vaginosis in non-pregnant women. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006055. doi: 10.1002/14651858.CD006055.pub2. PMID 19588379
- [Result] Joesoef MR, Schmid GP, Hillier SL. Bacterial vaginosis: review of treatment options and potential clinical indications for therapy. Clin Infect Dis. 1999 Jan;28 Suppl 1:S57-65. doi: 10.1086/514725. PMID 10028110
- [Result] Larsson PG, Carlsson B. Does pre- and postoperative metronidazole treatment lower vaginal cuff infection rate after abdominal hysterectomy among women with bacterial vaginosis? Infect Dis Obstet Gynecol. 2002;10(3):133-40. doi: 10.1155/S1064744902000133. PMID 12625969
- [Result] Larsson PG. Treatment of bacterial vaginosis. Int J STD AIDS. 1992 Jul-Aug;3(4):239-47. doi: 10.1177/095646249200300402. No abstract available. PMID 1504154
- [Result] McElligott KA, Havrilesky LJ, Myers ER. Preoperative screening strategies for bacterial vaginosis prior to elective hysterectomy: a cost comparison study. Am J Obstet Gynecol. 2011 Nov;205(5):500.e1-7. doi: 10.1016/j.ajog.2011.07.012. Epub 2011 Jul 20. PMID 21944221
- [Result] Schey D, Salom EM, Papadia A, Penalver M. Extensive fever workup produces low yield in determining infectious etiology. Am J Obstet Gynecol. 2005 May;192(5):1729-34. doi: 10.1016/j.ajog.2004.11.049. PMID 15902186
- [Result] Makinen J, Johansson J, Tomas C, Tomas E, Heinonen PK, Laatikainen T, Kauko M, Heikkinen AM, Sjoberg J. Morbidity of 10 110 hysterectomies by type of approach. Hum Reprod. 2001 Jul;16(7):1473-8. doi: 10.1093/humrep/16.7.1473. PMID 11425832
- [Result] Faro C, Faro S. Postoperative pelvic infections. Infect Dis Clin North Am. 2008 Dec;22(4):653-663. doi: 10.1016/j.idc.2008.05.005. PMID 18954757
- [Result] Lake AG, McPencow AM, Dick-Biascoechea MA, Martin DK, Erekson EA. Surgical site infection after hysterectomy. Am J Obstet Gynecol. 2013 Nov;209(5):490.e1-9. doi: 10.1016/j.ajog.2013.06.018. Epub 2013 Jun 13. PMID 23770467
- [Result] Tamussino K. Postoperative infection. Clin Obstet Gynecol. 2002 Jun;45(2):562-73. doi: 10.1097/00003081-200206000-00026. No abstract available. PMID 12048413
- [Result] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Result] American College of Obstetricians and Gynecologists Women's Health Care Physicians; Committee on Gynecologic Practice. Committee Opinion No. 571: Solutions for surgical preparation of the vagina. Obstet Gynecol. 2013 Sep;122(3):718-20. doi: 10.1097/01.AOG.0000433982.36184.95. PMID 23963423
- [Result] Lin L, Song J, Kimber N, Shott S, Tangora J, Aroutcheva A, Mazees MB, Wells A, Cohen A, Faro S. The role of bacterial vaginosis in infection after major gynecologic surgery. Infect Dis Obstet Gynecol. 1999;7(3):169-74. doi: 10.1002/(SICI)1098-0997(1999)7:33.0.CO;2-J. PMID 10371477
- [Result] Kenyon C, Colebunders R, Crucitti T. The global epidemiology of bacterial vaginosis: a systematic review. Am J Obstet Gynecol. 2013 Dec;209(6):505-23. doi: 10.1016/j.ajog.2013.05.006. Epub 2013 May 6. PMID 23659989
- [Result] Allsworth JE, Peipert JF. Prevalence of bacterial vaginosis: 2001-2004 National Health and Nutrition Examination Survey data. Obstet Gynecol. 2007 Jan;109(1):114-20. doi: 10.1097/01.AOG.0000247627.84791.91. PMID 17197596
- [Result] Koumans EH, Sternberg M, Bruce C, McQuillan G, Kendrick J, Sutton M, Markowitz LE. The prevalence of bacterial vaginosis in the United States, 2001-2004; associations with symptoms, sexual behaviors, and reproductive health. Sex Transm Dis. 2007 Nov;34(11):864-9. doi: 10.1097/OLQ.0b013e318074e565. PMID 17621244
- [Result] Fethers KA, Fairley CK, Hocking JS, Gurrin LC, Bradshaw CS. Sexual risk factors and bacterial vaginosis: a systematic review and meta-analysis. Clin Infect Dis. 2008 Dec 1;47(11):1426-35. doi: 10.1086/592974. PMID 18947329
- [Result] Esber A, Vicetti Miguel RD, Cherpes TL, Klebanoff MA, Gallo MF, Turner AN. Risk of Bacterial Vaginosis Among Women With Herpes Simplex Virus Type 2 Infection: A Systematic Review and Meta-analysis. J Infect Dis. 2015 Jul 1;212(1):8-17. doi: 10.1093/infdis/jiv017. Epub 2015 Jan 14. PMID 25589333
- [Result] Jamieson DJ, Duerr A, Klein RS, Paramsothy P, Brown W, Cu-Uvin S, Rompalo A, Sobel J. Longitudinal analysis of bacterial vaginosis: findings from the HIV epidemiology research study. Obstet Gynecol. 2001 Oct;98(4):656-63. doi: 10.1016/s0029-7844(01)01525-3. PMID 11576584
- [Result] Yen S, Shafer MA, Moncada J, Campbell CJ, Flinn SD, Boyer CB. Bacterial vaginosis in sexually experienced and non-sexually experienced young women entering the military. Obstet Gynecol. 2003 Nov;102(5 Pt 1):927-33. doi: 10.1016/s0029-7844(03)00858-5. PMID 14672465
- [Result] Klebanoff MA, Schwebke JR, Zhang J, Nansel TR, Yu KF, Andrews WW. Vulvovaginal symptoms in women with bacterial vaginosis. Obstet Gynecol. 2004 Aug;104(2):267-72. doi: 10.1097/01.AOG.0000134783.98382.b0. PMID 15291998
- [Result] Goldenberg RL, Klebanoff MA, Nugent R, Krohn MA, Hillier S, Andrews WW. Bacterial colonization of the vagina during pregnancy in four ethnic groups. Vaginal Infections and Prematurity Study Group. Am J Obstet Gynecol. 1996 May;174(5):1618-21. doi: 10.1016/s0002-9378(96)70617-8. PMID 9065140
- [Result] Amsel R, Totten PA, Spiegel CA, Chen KC, Eschenbach D, Holmes KK. Nonspecific vaginitis. Diagnostic criteria and microbial and epidemiologic associations. Am J Med. 1983 Jan;74(1):14-22. doi: 10.1016/0002-9343(83)91112-9. PMID 6600371
- [Result] Workowski KA, Bolan GA; Centers for Disease Control and Prevention. Sexually transmitted diseases treatment guidelines, 2015. MMWR Recomm Rep. 2015 Jun 5;64(RR-03):1-137. PMID 26042815
- [Result] Landers DV, Wiesenfeld HC, Heine RP, Krohn MA, Hillier SL. Predictive value of the clinical diagnosis of lower genital tract infection in women. Am J Obstet Gynecol. 2004 Apr;190(4):1004-10. doi: 10.1016/j.ajog.2004.02.015. PMID 15118630
- [Result] Al-Banna NA, Pavlovic D, Grundling M, Zhou J, Kelly M, Whynot S, Hung O, Johnston B, Issekutz TB, Kern H, Cerny V, Lehmann Ch. Impact of antibiotics on the microcirculation in local and systemic inflammation. Clin Hemorheol Microcirc. 2013;53(1-2):155-69. doi: 10.3233/CH-2012-1583. PMID 22975936
- [Result] Thulkar J, Kriplani A, Agarwal N. A comparative study of oral single dose of metronidazole, tinidazole, secnidazole and ornidazole in bacterial vaginosis. Indian J Pharmacol. 2012 Mar;44(2):243-5. doi: 10.4103/0253-7613.93859. PMID 22529484
- [Result] Austin MN, Beigi RH, Meyn LA, Hillier SL. Microbiologic response to treatment of bacterial vaginosis with topical clindamycin or metronidazole. J Clin Microbiol. 2005 Sep;43(9):4492-7. doi: 10.1128/JCM.43.9.4492-4497.2005. PMID 16145097
- [Result] Lugo-Miro VI, Green M, Mazur L. Comparison of different metronidazole therapeutic regimens for bacterial vaginosis. A meta-analysis. JAMA. 1992 Jul 1;268(1):92-5. PMID 1535108
- [Derived] Lopez CC, Villegas-Echeverri JD, De Los Rios JF, Vasquez-Trespalacios EM, Arango A, Cifuentes C, Orjuela J, Valencia V, Cardenas L, Lopez JD, Lopez JD, Zambrano CP, Gomez SM, Bastidas C, Silva JB, Gallego DE. Metronidazole for Prevention of Pelvic Cellulitis and Abscess after Laparoscopic Hysterectomy: A Triple-blinded, Randomized, Placebo-controlled Clinical Trial. J Minim Invasive Gynecol. 2023 Nov;30(11):912-918. doi: 10.1016/j.jmig.2023.07.007. Epub 2023 Jul 16. PMID 37463650